CLINICAL TRIAL: NCT04332198
Title: Neurobiological and Neuro-immunological Mechanisms of Dyspnea in Amyotrophic Lateral Sclerosis
Brief Title: Neurobiological and Immunological Mechanisms of Dyspnea in ALS (BIOPNEA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Association pour le Développement et l'Organisation de la Recherche en Pneumologie et sur le Sommeil (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019_A02882_55
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Shortness of Breath; Dyspnea; Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Dyspnea; Amyotrophic Lateral Sclerosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ALS patients (Experimental)
  Interventions: Other: biological test

INTERVENTIONS:
Other: biological test — dyspnea evaluation, ventilatory evaluation and biological test before and after non invasive ventilation
  Other Names: questionnaire

SUMMARY:
Dyspnea; subjective experience of respiratory discomfort; which produces negative emotional experience, is the most common symptom of patients afflicted with chronic respiratory failure and its treatments are limited. Amyotrophic Lateral Sclerosis (ALS) related - dyspnea, due to diaphragmatic dysfunction, is similar to dyspnea during mechanical inspiratory load (activation of the supplementary motor area, SMA). The perception of pain and dyspnea is processed in similar brain areas (insula, dorsal anterior cingulate cortex, amygdala and medial thalamus) and in ALS; relieving dyspnea by noninvasive ventilation (NIV) is associated with decreased pain thresholds. Otherwise, it is reported systemic elevations of pro-inflammatory cytokines in chronic pain patients, correlating with intensity of pain, and during respiratory load in healthy volunteers.

The objectives are to evaluate the cytokines and endorphins rates variations after initiation of NIV in ALS patients, and to correlate cytokines and endorphins rates with the intensity of the affective component and the intensity of the sensory component of dyspnea.

The investigators will perform a prospective, experimental study, including 30 ALS patients. Dyspnea, ventilatory and cardiac settings, electromyographic recording of the scalene muscle and biological assays (ACTH, endorphin, Neuropeptide P, BDNF, IL1, IL6, IL8, IL10, TNF), will be measured during spontaneous breathing and during NIV at different times after initiation.

The investigators expect a reduction of immunological and neurobiological markers after relieving dyspnea by NIV. This work could lead to the development of new treatments for dyspnea.

ELIGIBILITY:
Inclusion Criteria:

- Patients with chronic respiratory failure with diaphragmatic dysfunction linked to amyotrophic lateral sclerosis and requiring long-term NIV

Exclusion Criteria:

* Other respiratory disease (COPD, asthma, obstructive sleep apnea)
* Alcohol or psychotropic drug the lasts 24 hours
* Cognitive impairment
* Smoking > 10 PA
* Exacerbation or infection 6 weeks earlier
* Endstage of illness
* Chronic or acute pain (VAS > 3)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
the cytokines and endorphins rates variation after initiation of NIV in ALS patients | 30 minutes
  measure cytokines and endorphins blood levels before and after NIV